CLINICAL TRIAL: NCT00486330
Title: Pharmacokinetic Interactions Between Buprenorphine/Naloxone and Tipranavir/Ritonavir in HIV-Negative Subjects Chronically Receiving Buprenorphine/Naloxone
Brief Title: Pharmacokinetic Interactions Between Buprenorphine and Tipranavir/Ritonavir
Acronym: BUTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, R. Douglas Bruce, MD, MA, Principal Investigator, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0505027698
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: HIV Infections
Keywords: HIV; Pharmacokinetics; Buprenorphine; Tipranavir; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Buprenorphine; tipranavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Buprenorphine plus Tipranavir/Ritonavir (Other)
  Interventions: Drug: Buprenorphine, Tipranavir and ritonavir

INTERVENTIONS:
Drug: Buprenorphine, Tipranavir and ritonavir — After determining buprenorphine/naloxone pharmacokinetics over a 24-hour period, tipranavir/ritonavir and buprenorphine/naloxone will be coadministered for 7 days.

SUMMARY:
The main purpose of this study is to examine the effect of tipranavir combined with ritonavir, medications for the treatment of HIV-infection, on buprenorphine/naloxone (BUP) in people who have been receiving the same dose of buprenorphine/naloxone for at least 3 weeks before study entry.

DETAILED DESCRIPTION:
A large number of people with HIV-infection obtained HIV through injection drug use. Some of these people are currently being treated with buprenorphine/naloxone (BUP) for their addiction and with medications for HIV infection. Tipranavir is a medication that was recently approved by the Food and Drug Administration (FDA) for the treatment of HIV-infection. Tipranavir is given in combination with another HIV medication, ritonavir. Tipranavir acts by making it more difficult for the virus that causes AIDS to multiply and cause more damage to the immune system. Ritonavir acts by increasing the amount of tipranavir available to fight HIV.

Earlier studies looking at the combination of BUP and HIV medications have shown that BUP and some HIV medications act differently when taken together. It is important to learn if taking BUP and HIV medications together results in changes in the blood level of either medication. If the HIV medication decreases the level of BUP in the blood, an individual taking BUP and HIV medications may experience symptoms of withdrawal ("dope sickness"), even while taking their usual dose of BUP. On the other hand, if BUP decreases the amount of HIV medication in the blood, then the HIV medication may be less effective in controlling HIV infection. It is therefore important to learn if tipranavir/ritonavir and BUP will affect each other when taken together.

In order to learn about the effects of BUP on tipranavir/ritonavir, we will need to measure the amount of BUP in your blood for 24 hours after you have taken tipranavir/ritonavir and BUP together and then compare that to the amount of BUP in your blood when you are not taking tipranavir/ritonavir.

ELIGIBILITY:
Inclusion Criteria:

* Buprenorphine/naloxone (BUP/NAL) users (taking 16/4 mg sublingually daily) for at least 3 weeks deemed by the investigator to have acceptable medical history, physical examination, 12 lead electrocardiogram, and clinical laboratory evaluations consistent with BUP maintenance will be eligible to participate in the study.
* Subjects who meet the criteria of opiate dependence, are enrolled in long-term BUP maintenance therapy, and have been on a stable dose of BUP/NAL for at least 3 weeks.
* Body weight > 60 kg for males and > 40 kg for females
* Body Mass Index (BMI) of 18 to 30 kg/m2, inclusive. BMI = weight (kg)/ [height(m)]2.
* Male or females, ages > 18 to < 60 years.
* Women of childbearing potential (WOCBP) must not be nursing or pregnant and must be on adequate non-hormonal contraception to avoid pregnancy. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of Study Day 1.

Exclusion Criteria:

* History or current evidence of any significant acute or chronic medical illness that, within the investigator's discretion, would interfere with the conduct or interpretation of the study.
* History of acute or chronic pancreatitis.
* History of uncontrolled chronic medical illness which could adversely affect the subject's adherence to study protocol or affect patient safety in the opinion of the investigator
* Use of any medication thought to significantly alter the metabolism of tipranavir, ritonavir, Buprenorphine or naloxone.
* History of any hemolytic disorders (including drug-induced hemolysis).
* Proven or suspected acute hepatitis at the time of study entry.
* Chronic liver disease with Childs-Pugh Class B or C staging
* Current or recent (within 3 months) gastrointestinal disease which would interfere with the conduct or interpretation of the study.
* Any major surgery within 4 weeks of enrollment. Minor surgical procedures requiring local anesthesia are exceptions.
* Any gastrointestinal surgery that could impact upon the absorption of study drug.
* Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks of enrollment.
* Blood transfusion within 4 weeks of enrollment.
* Inability to tolerate oral medication.
* Inability to tolerate venipuncture and/or absence of secure venous access.
* Inability to refrain from smoking during in-residence period
* Known or suspected HIV infection (subjects who are found to be positive upon screen for HIV will be excluded).
* Known active drug or alcohol abuse, which in the opinion of the investigator makes study participation to completion unlikely.
* Any other sound medical, psychiatric and/or social reason as determined by the Investigator.
* Evidence of organ dysfunction or any clinically relevant (as determined by the investigator) deviations from the norms observed in a buprenorphine/naloxone treated population in physical examination, vital signs, ECG or clinical laboratory determinations.
* Ingestion of alcohol within 24 hours prior to the dose of study medication
* Positive breathalyzer alcohol test, or positive urine screen for barbiturates, benzo-diazepines, amphetamines, THC, cocaine or opiates other than buprenorphine/naloxone.
* Positive blood screen for HIV antibody.
* Subjects with AST, ALT or bilirubin > 2.5X the upper limit of normal.
* Hemoglobin < 9 g/dL, and platelet count < 75, 000/mm3.
* Positive serum or urine for HCG.
* History of any significant drug allergy, drug rash or sensitivity to any class of drugs relevant to the study drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Bruce, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine AIDS Program, New Haven, Connecticut, United States

REFERENCES:
- [Result] Bruce RD, Altice FL, Moody DE, Lin SN, Fang WB, Sabo JP, Wruck JM, Piliero PJ, Conner C, Andrews L, Friedland GH. Pharmacokinetic interactions between buprenorphine/naloxone and tipranavir/ritonavir in HIV-negative subjects chronically receiving buprenorphine/naloxone. Drug Alcohol Depend. 2009 Dec 1;105(3):234-9. doi: 10.1016/j.drugalcdep.2009.07.007. Epub 2009 Sep 1. PMID 19726139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from buprenorphine maintenance treatment in New Haven over a year period. Subjects were hospitalized at baseline to be stabilized on buprenorphine/naloxone (BUP/NLX) therapy.
Pre-assignment Details: There were no pre-assignment exclusion criteria.
Groups:
- Tipranavir/Ritonavir (500mg/200mg): Subjects on buprenorphine maintenance therapy prior to starting the study. Subsequently, tipranavir 500 mg and ritonavir 200 mg (TPV/r) was administered twice daily for a minimum of 7 days. Subjects served as their own controls. PK parameters were evaluated Pre- and Post-administration of tipranavir.
Period: Overall Study
Arm/Group | Tipranavir/Ritonavir (500mg/200mg)
Started | 12 (Twelve subjects met inclusion/exclusion criteria)
Completed | 10 (Of the 12 subjects treated, two developed adverse events leading to study drug discontinuation.)
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tipranavir/Ritonavir (500mg/200mg)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 44 (10) [21 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of BUP/NLX With TPV/r (h*ng/mL)
Description: Non-compartmental methods were used for pharmacokinetic analysis. The area under the plasma drug concentration-time curve was estimated by linear-log trapezoidal rule at 24-hrs.
Time Frame: 10 days
Measure: Geometric Mean (Full Range); unit: h*ng/mL
Groups:
- Tipranavir/Ritonavir (500mg/200mg): Subjects on buprenorphine maintenance therapy prior to starting the study. Subsequently, tipranavir 500 mg and ritonavir 200 mg was administered twice daily for a minimum of 7 days. Subjects served as their own controls. PK parameters were evaluated Pre- and Post-administration of tipranavir.
Arm/Group | Tipranavir/Ritonavir (500mg/200mg)
Number analyzed (Participants) | 10
h*ng/mL | 43.7 [16.4 to 112.7]

ADVERSE EVENTS:
Arm/Group | Tipranavir/Ritonavir (500mg/200mg)
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tipranavir/Ritonavir (500mg/200mg) (N=12)
Elevated transaminases (Hepatobiliary disorders) | 1 (1) — one subject withdrew due to elevated hepatic transaminases (>5x ULN; DAIDS Grade 3) detected during routine screening on day 4 which was attributed to known hepatic effects of tipranavir (2005).
Perioral numbness and lightheadedness (Nervous system disorders) | 1 (1) — One subject withdrew due to perioral numbness and lightheadedness likely due to RTV after the first day of study drug administration (Ritonavir Package Insert 2007)

LIMITATIONS AND CAVEATS:
First, the sample size was small. Second, this study utilized a within-subject design with patients acting as their own controls and thereby resulting in less intra-patient variability in the analysis of BUP/NLX.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No